CLINICAL TRIAL: NCT00919503
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Nonmalignant Inherited Disorders Using a Treosulfan Based Preparative Regimen
Brief Title: Treosulfan and Fludarabine Phosphate Before Donor Stem Cell Transplant in Treating Patients With Nonmalignant Inherited Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: medac GmbH (Industry); National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lauri Burroughs, Associate Professor, Clinical Research Division, Fred Hutch; Director, Non-Malignant Transplant Program, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2256.00; NCI-2010-01277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2256.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG2809001 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Non-Neoplastic Hematologic and Lymphocytic Disorder
Keywords: nonmalignant diseases; nonmalignant inherited disorders; primary immunodeficiency diseases; primary immune deficiency disorders; chronic granulomatous; disease; IPEX syndrome; hemophagocytic lymphohistiocytosis; Wiskott Aldrich Syndrome; bone marrow failure syndromes; Shwachman Diamond Syndrome; Dyskeratosis Congenita; Diamond Blackfan Anemia; inborn errors of metabolism; metabolic diseases; hemoglobinopathies; sickle cell disease; thalassemia; reduced intensity transplantation; hematopoietic cell transplantation; bone marrow transplantation; umbilical cord blood transplantation
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Disease; Immune Dysregulation, Polyendocrinopathy, Enteropathy, X-Linked Syndrome; Lymphohistiocytosis, Hemophagocytic; Wiskott-Aldrich Syndrome; Bone Marrow Failure Disorders; Shwachman-Diamond Syndrome; Dyskeratosis Congenita; Anemia, Diamond-Blackfan; Metabolism, Inborn Errors; Metabolic Diseases; Hemoglobinopathies; Anemia, Sickle Cell; Thalassemia | interventions — Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; fludarabine phosphate; Methotrexate; merphos; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation; treosulfan; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Regimen A (PBSCT and BMT) (Experimental): CONDITIONING REGIMEN A : Patients receive treosulfan IV on days -6 to -4 and fludarabine phosphate IV on days -6 to -2. Patients receive anti-thymocyte globulin IV on days -4 to -2. Patients undergoing umbilical cord blood transplantation will also receive low dose total-body irradiation on day -1.
  TRANSPLANTATION: Patients receive either bone marrow, peripheral blood stem cells (PBSC), or umbilical cord blood from the donor on day 0. The use of either bone marrow, PBSC, or umbilical cord blood will depend on the donor status.
  Patients undergoing bone marrow or PBSC transplantation receive tacrolimus IV continuously or PO twice daily on days -1 to 50 followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Drug: Treosulfan
- Regimen B (UBCT) (Experimental): CONDITIONING REGIMEN B: Patients receive treosulfan IV on days -6 to -4 and fludarabine phosphate IV on days -6 to -2. Patients receive anti-thymocyte globulin IV on days -4 to -2. Patients undergoing umbilical cord blood transplantation will also receive low dose total-body irradiation on day -1 .
  TRANSPLANTATION: Patients receive either bone marrow, peripheral blood stem cells (PBSC), or umbilical cord blood from the donor on day 0. The use of either bone marrow, PBSC, or umbilical cord blood will depend on the donor status.
  Patients undergoing UCB transplantation receive cyclosporine IV over 1 hour every 8-12 hours on days -3 to 100 followed by a taper until day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil IV or PO every 8 hours on days 0 to 40 followed by a taper until day 96 in the absence of GVHD.
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Drug: Treosulfan; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Infused IV
  Other Names: Allo BMT; Allogeneic BMT
  Arms: Regimen A (PBSCT and BMT)
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Cyclosporine — Given IV or PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
  Arms: Regimen B (UBCT)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Regimen A (PBSCT and BMT)
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
  Arms: Regimen B (UBCT)
Procedure: Peripheral Blood Stem Cell Transplantation — Infused IV
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
  Arms: Regimen A (PBSCT and BMT)
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
  Arms: Regimen A (PBSCT and BMT)
Radiation: Total-Body Irradiation — Undergo total body irradiation
  Other Names: Total Body Irradiation; Whole-Body Irradiation
  Arms: Regimen B (UBCT)
Drug: Treosulfan — Given IV
  Other Names: 1,2,3, 4-Butanetetrol, 1,4-dimethanesulfonate, [R-(R*,S*)]-; Dihydroxybusulfan; Ovastat; Treosulphan; Tresulfon
Procedure: Umbilical Cord Blood Transplantation — Single or double unit umbilical cord blood transplant, infused IV
  Other Names: Cord Blood Transplantation; UCB transplantation
  Arms: Regimen B (UBCT)

SUMMARY:
This phase II clinical trial studies how well treosulfan and fludarabine phosphate with or without low dose radiation before donor stem cell transplantation works in treating patients with nonmalignant (noncancerous) diseases. Hematopoietic cell transplantation has been shown to be curative for many patients with nonmalignant (noncancerous) diseases such as primary immunodeficiency disorders, bone marrow failure syndromes, hemoglobinopathies, and inborn errors of metabolism (metabolic disorders). Powerful chemotherapy drugs and/or radiation are often used to condition the patient before infusion of the new healthy donor cells. The purpose of the conditioning therapy is to destroy the patient's abnormal bone marrow which doesn't work properly in order to make way for the new healthy donor cells which functions normally. Although effective in curing the patient's disease, many hematopoietic cell transplantation regimens use intensive chemotherapy and/or radiation which can be quite toxic, have significant side effects, and can potentially be life-threatening. Investigators are investigating whether a new conditioning regimen that uses less intensive drugs (treosulfan and fludarabine phosphate) with or without low dose radiation results in new blood-forming cells (engraftment) of the new donor cells without increased toxicities in patients with nonmalignant (noncancerous) diseases.

DETAILED DESCRIPTION:
OUTLINE:

CONDITIONING REGIMEN: Patients receive treosulfan intravenously (IV) over 2 hours on days -6 to -4 and fludarabine phosphate IV over 1 hour on days -6 to -2. Patients receive anti-thymocyte globulin IV over 4-6 hours on days -4 to -2. Patients undergoing umbilical cord blood transplantation will also receive low dose total-body irradiation on day -1.

TRANSPLANTATION: Patients receive either bone marrow, peripheral blood stem cells (PBSC), or umbilical cord blood (UCB) from the donor on day 0. The use of either bone marrow, PBSC, or umbilical cord blood will depend on the donor status.

IMMUNOSUPPRESSION: Patients receive a combination of immunosuppressive medications to try and prevent graft-versus-host disease. There are 2 regimens depending on the donor.

Regimen A: Patients undergoing bone marrow or PBSC transplantation receive tacrolimus daily from day -1 to 50 followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Regimen B: Patients undergoing UCB transplantation receive cyclosporine on days -3 to 100 followed by a taper until day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil on days 0 to 40 followed by a taper until day 96 in the absence of GVHD.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a nonmalignant disease treatable by allogeneic HCT
* Patients with a known nonmalignant disease that is not clearly defined will need to be discussed with the protocol principal investigator (PI) (Dr. Lauri Burroughs) and potentially the nonmalignant board to determine if they are eligible for HCT on this study
* DONOR: Human leukocyte antigens (HLA)-identical related donors or unrelated donors matched for HLA-A, B, C, DRB1, and DQB1 or mismatched for a single allele at HLA-A, B, C, DRB1 or a single DQB1 antigen or allele mismatch by high resolution deoxyribonucleic acid (DNA) typing
* DONOR: PBSC is the preferred cell source (when feasible) for fully matched donors; PBSC may also be used for a mismatched donor following discussion with the PI; bone marrow is allowed when PBSC is not feasible or as determined by the PI
* DONOR: HLA-matched sibling bone marrow in combination with HLA-matched sibling umbilical cord blood if the HLA-matched sibling umbilical cord blood was collected and stored; the HLA-matched sibling bone marrow and cord blood would be matched for HLA-A, B, C, DRB1, and DQB1
* DONOR: Unrelated Umbilical Cord Blood: Unit selection is based on the cryopreserved total nucleated cell (TNC) dose and matching at HLA-A, B antigen level and DRB1 allele level typing; while HLA-C antigen/allele level typing is not considered in the matching criteria, if available, may be used to optimize unit selection
* DONOR: Unrelated Umbilical Cord Blood: The patient and the cord blood unit(s) must be matched for at least 4 of 6 loci as defined above
* DONOR: Unrelated Umbilical Cord Blood: Selection of two umbilical cord blood (UCB) units is allowed to provide sufficient cell dose
* DONOR: Unrelated Umbilical Cord Blood: The UCB unit with the least HLA disparity (with the patient) will be selected first (i.e., selection priority is 6/6 match > 5/6 match> 4/6 match); additional UCB units then may be selected to achieve the required cell dose; if a second unit is required, this unit will be the unit that most closely HLA matches the patient and meets minimum size criteria outlined below of at least 1.5 x 10^7 TNC/kg (i.e. a smaller more closely matched unit will be selected over a larger less well matched unit as long as minimum criteria are met)
* DONOR: Unrelated Umbilical Cord Blood: Each UCB unit MUST contain at least 1.5 x 10^7 TNC per kilogram recipient weight
* DONOR: Unrelated Umbilical Cord Blood: The total cell dose of the combined units must be at least 3.0 x 10^7 TNC per kilogram recipient weight

Exclusion Criteria:

* Patients with idiopathic aplastic anemia and Fanconi anemia; (patients with aplastic anemia associated with paroxysmal nocturnal hemoglobinuria [PNH] or inherited marrow failure syndromes, except Fanconi anemia, will be allowed)
* Patients with impaired cardiac function as evidenced by ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%) or cardiac insufficiency requiring treatment or symptomatic coronary artery disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Patients with impaired pulmonary function as evidenced by diffusion capacity of the lung for carbon monoxide (DLCO) < 50% of predicted (or, if unable to perform pulmonary function tests, then oxygen [O2] saturation < 92% on room air)
* Patients with impaired renal function as evidenced by creatinine-clearance < 50% for age, weight, height or serum creatinine > 2 x upper normal limit or dialysis-dependent
* Patients with evidence of synthetic dysfunction or severe cirrhosis requiring deferral of conditioning as recommended by a gastroenterology specialist
* Patients with an active infectious disease requiring deferral of conditioning; as recommended by an infectious disease specialist
* Patients who are positive for human immunodeficiency virus (HIV)
* Females who are pregnant or breast-feeding
* Patients with a known hypersensitivity to treosulfan and/or fludarabine
* Receiving another experimental drug within 4 weeks of initiation of conditioning (day -6) unless approved by the PI
* DONOR: Deemed unable to undergo marrow harvesting or PBSC mobilization and leukapheresis
* DONOR: HIV-positive
* DONOR: With active infectious hepatitis
* DONOR: Females with a positive pregnancy test
* DONOR: HLA-matched sibling cord blood exclusions: Any cord blood units that have not passed donor screening for infectious disease markers as recommended by the National Marrow Donor Project (NMDP) will not be used unless a waiver is signed by the clinical attending allowing use of cord blood unit; cord blood units are presumed to be cytomegalovirus (CMV) negative regardless of serologic testing due to passive transmission of maternal CMV antibodies
* DONOR: Unrelated Umbilical Cord Blood: Any cord blood units with < 1.5 x 10^7 total nucleated cells per kilogram recipient weight
* DONOR: Unrelated Umbilical Cord Blood: Any cord blood units that have not passed donor screening for infectious disease markers as recommended by NMDP will not be used unless a waiver is signed by the clinical attending allowing use of cord blood unit; cord blood units are presumed to be CMV negative regardless of serologic testing due to passive transmission of maternal CMV antibodies

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauri M. Burroughs, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A (PBSCT and BMT): CONDITIONING REGIMEN A : Patients receive treosulfan IV on days -6 to -4 and fludarabine phosphate IV on days -6 to -2. Patients receive anti-thymocyte globulin IV on days -4 to -2. Patients undergoing umbilical cord blood transplantation will also receive low dose total-body irradiation on day -1.
  TRANSPLANTATION: Patients receive either bone marrow, peripheral blood stem cells (PBSC), or umbilical cord blood from the donor on day 0. The use of either bone marrow, PBSC, or umbilical cord blood will depend on the donor status.
  Patients undergoing bone marrow or PBSC transplantation receive tacrolimus IV continuously or PO twice daily on days -1 to 50 followed by a taper until day 180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Allogeneic Bone Marrow Transplantation: Infused IV
  Anti-Thymocyte Globulin: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IV
  Peripheral Blood Stem Cell Transplantation: Infused IV
  Tacrolimus: Given IV or PO
  Treosulfan: Given IV
- Regimen B (UBCT): CONDITIONING REGIMEN B: Patients receive treosulfan IV on days -6 to -4 and fludarabine phosphate IV on days -6 to -2. Patients receive anti-thymocyte globulin IV on days -4 to -2. Patients undergoing umbilical cord blood transplantation will also receive low dose total-body irradiation on day -1 .
  TRANSPLANTATION: Patients receive either bone marrow, peripheral blood stem cells (PBSC), or umbilical cord blood from the donor on day 0. The use of either bone marrow, PBSC, or umbilical cord blood will depend on the donor status.
  Patients undergoing UCB transplantation receive cyclosporine IV over 1 hour every 8-12 hours on days -3 to 100 followed by a taper until day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil IV or PO every 8 hours on days 0 to 40 followed by a taper until day 96 in the absence of GVHD.
  Anti-Thymocyte Globulin: Given IV
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Total-Body Irradiation: Undergo total body irradiation
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation: Single or double unit umbilical cord blood transplant, infused IV
Period: Overall Study
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Started | 84 | 14
Completed | 84 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT) | Total
Number analyzed (Participants) | 84 | 14 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70 | 13 | 83
  Between 18 and 65 years | 14 | 1 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 3 | 31
  Male | 56 | 11 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 77 | 10 | 87
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 1 | 9
  White | 67 | 9 | 76
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 84 | 14 | 98

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Efficacy
Description: Number of patients engrafted (>5% donor CD3+ peripheral blood chimerisms) at 1 year following transplant
Time Frame: 1 year following transplant
Population: Regimen B: Three patients expired without CD3+ chimerisms being performed, therefore could not be analyzed for primary efficacy
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 11
Participants | 83 | 10

2. Secondary Outcome: Non-relapse Mortality
Description: Number of patients who experienced non-relapse mortality by 1 year following transplant
Time Frame: 1 year following transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 14
Participants | 2 | 5

3. Secondary Outcome: Number of Patients With Grade II-IV Acute Graft-versus-host Disease
Description: Number of patients diagnosed with overall grade II-IV acute GVHD by Day 100 post transplant
Time Frame: Day 100 post transplant
Population: Regimen B: 2 patients expired too early for evaluation for acute GVHD and could not be evaluated for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 12
Participants | 44 | 8

4. Secondary Outcome: Number of Patients With of Chronic Graft-versus-host Disease
Description: Number of patients diagnosed with chronic GVHD and requiring systemic immunosuppression within 1 year following transplant
Time Frame: 1 year following transplant
Population: Regimen B: 3 patients expired too early for evaluation for chronic GVHD and could not be evaluated for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 11
Participants | 29 | 5

5. Secondary Outcome: Donor Chimerism CD3 at 100 Days Post Transplant
Description: Number of patients with peripheral blood donor chimerism for CD3 less than 5%, 5-49%, 50-94% and greater than or equal to 95% at 100 days post transplant.
Time Frame: Day 100 post transplant
Population: Regimen B: 3 patients expired without CD3+ chimerisms being performed and could not be evaluated for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 11
Participants
  Greater than equal to 95% | 49 | 7
  50 - 94% | 29 | 2
  5-49% | 6 | 1
  Less than 5% | 0 | 1

6. Secondary Outcome: Disease Response at One Year Following Hematopoietic Cell Transplantation
Description: Number of patients with no evidence of disease at one year following transplant
Time Frame: 1 year following transplant
Population: Regimen B: 3 patients expired prior to disease response being evaluated and could not be evaluated for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 11
Participants | 78 | 8

7. Secondary Outcome: Immune Reconstitution Following Hematopoietic Cell Transplantation
Description: Number of patients with immune reconstitution (defined by a normal range CD3) at 1 year post transplant
Time Frame: 1 year following transplant
Population: Regimen A: 11 patients did not have lymphocyte subsets drawn post-transplant and could not be evaluated for outcome; Regimen B: 3 patients expired prior to lymphocyte subsets being evaluated and 2 patients did not have lymphocyte subsets drawn post-transplant and could not be evaluated for outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 73 | 9
Participants | 39 | 4

8. Secondary Outcome: Number of Participants With Infections
Description: Number of participants with clinically significant infections (bacterial, fungal, viral) requiring treatment within 100 days following transplant
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 14
Participants | 57 | 9

9. Secondary Outcome: Overall Survival
Description: Number of patients alive at 1 year following transplant
Time Frame: 1 year following transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 14
Participants | 80 | 9

10. Secondary Outcome: Donor Chimerism CD33 at Day 100 Post Transplant
Description: Number of patients with peripheral blood donor chimerism for CD33 less than 5%, 5-49%, 50-94% and greater than or equal to 95% at 100 days post transplant.
Time Frame: 100 days post transplant
Population: Regimen B: 2 patients expired without CD33+ chimerisms being performed and could not be evaluated for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
Number analyzed (Participants) | 84 | 12
Participants
  Greater than equal to 95% | 72 | 7
  50-94% | 8 | 2
  5-49% | 4 | 2
  Less than 5% | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 100 post initiation of conditioning therapy
Description: Adverse Events were collected 100 days post initiation of conditioning therapy. All-Cause Mortality was assessed through 10.6 years post transplant (through study completion date 6/10/2020).
Arm/Group | Regimen A (PBSCT and BMT) | Regimen B (UBCT)
All-Cause Mortality (participants affected / at risk) | 7/84 | 6/14
Serious Adverse Events (participants affected / at risk) | 17/84 | 5/14
Other Adverse Events (participants affected / at risk) | 53/84 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (PBSCT and BMT) (N=84) | Regimen B (UBCT) (N=14)
Gastrointestinal Other: Pneumatosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — grade 4
Sepsis with multiorgan failure (Infections and infestations) | 0 (0) | 2 (2) — grade 5
Apnea: Requiring intubation following BAL; attributed to underlying infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — grade 4
Anaphylaxis reaction (rATG) (Immune system disorders) | 2 (2) | 0 (0) — grade 4
Cardiac Asystole following central venous catheter placement (Cardiac disorders) | 1 (1) | 0 (0) — grade 5
Hypotension: requiring intervention (Vascular disorders) | 1 (1) | 0 (0) — grade 3
Hypotension: shock, pressors (Vascular disorders) | 1 (1) | 0 (0) — grade 4
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) — grade 3
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3
Diarrhea (associated with GVHD): >15ml/kg per day with abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — grade 3
Fever (not neutropenic): attributed to rATG (General disorders) | 2 (2) | 0 (0) — grade 3
Fever (not neutropenic) (General disorders) | 2 (2) | 0 (0) — grade 3
Febrile neutropenia: attributed to rATG (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — grade 3
Febrile Neutropenia: with life- threatening sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — grade 4
Infections and infestations -Other, specify: parainfluenza or sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations -Other, specify: CMV meningitis/encephalo (Infections and infestations) | 1 (1) | 0 (0) — grade 3
Infections and infestations -Other, specify: Clostridium septicum sepsis (Infections and infestations) | 1 (1) | 0 (0) — grade 3
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — grade 4
Acute kidney injury (reversible, requiring CRRT/dialysis) (Renal and urinary disorders) | 1 (1) | 0 (0) — grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — grade 3
Hypoxia: Decreased O2 sat requiring support (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) — grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (PBSCT and BMT) (N=84) | Regimen B (UBCT) (N=14)
Anaphylaxis reaction: Possible reaction to rATG (Immune system disorders) | 1 (1) | 1 (1) — grade 3
Pericardial effusion: Tamponade (Cardiac disorders) | 0 (0) | 2 (3) — grade 4
Thrombotic microangiopathy (requiring intervention) with acute renal fail: Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — grade 4
Fluid retention - evidence of ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 3
Diarrhea (associated with GVHD): >15ml/kg per day (Gastrointestinal disorders) | 1 (1) | 1 (1) — grade 3
Gastrointestinal disorders -Other, specify: pneumatosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 3
Oral mucositis: Requiring intervention (Gastrointestinal disorders) | 20 (20) | 1 (1) — grade 3
Esophageal ulcers: Presumed viral esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — grade 3
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — grade 3
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — grade 3
Elevated bilirubin (>3-10x ULN) (Investigations) | 2 (2) | 2 (2) — grade 3
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (17) | 4 (4) — grade 3
Fever (not neutropenic): attributed to rATG (General disorders) | 6 (6) | 1 (1) — grade 3
Fever (not neutropenic) (General disorders) | 0 (0) | 1 (1) — grade 3
Infections and infestations -Other, specify: life-threatening disseminated Adenovirus (Infections and infestations) | 0 (0) | 1 (1) — grade 4
sleep apnea: Obstructive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — grade 3
Hypoxia: decreased O2 sat (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1) — grade 3
Hypoxia: requiring intubation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) — grade 4
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — grade 4
Acute kidney injury (reversible, requiring CRRT/dialysis) (Renal and urinary disorders) | 1 (1) | 1 (1) — grade 3
Hemolysis (AIHA): Requiring transfusion and sterioids (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — grade 3
Hypotension: requiring intervention (Vascular disorders) | 3 (3) | 0 (0) — grade 3
Cardiopulmonary arrest: Requiring intubation (Cardiac disorders) | 1 (1) | 0 (0) — grade 4
Thrombotic microangiopathy (not requiring intervention) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — grade 3
Rash (>50%) (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — grade 3
Colitis: Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) — grade 3
Febrile neutropenia: attributed to rATG (Blood and lymphatic system disorders) | 7 (7) | 0 (0) — grade 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — grade 3
Dysfunctional urerine (menstrual) bleeding: requiring transfusion (Reproductive system and breast disorders) | 1 (1) | 0 (0) — grade 3
Oral hemorrhage: Bleeding (requiring transfusion) (Gastrointestinal disorders) | 1 (1) | 0 (0) — grade 3
nfections and infestations -Other, specify: MSSA septic shock (Infections and infestations) | 1 (1) | 0 (0) — grade 4
Infections and infestations -Other, specify: Strep viridans, enterococcus bacteremia (Infections and infestations) | 1 (1) | 0 (0) — grade 3
Reversible posterior leukoencephalopathy syndrome (PRES) (Nervous system disorders) | 1 (1) | 0 (0) — grade 3
Seizure (conciousness altered) (Nervous system disorders) | 3 (5) | 0 (0) — grade 3
Carbon monoxide diffusing capacity decreased (DLCO) (Investigations) | 1 (1) | 0 (0) — grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT00919503/Prot_SAP_000.pdf